CLINICAL TRIAL: NCT04151810
Title: Phase I Clinical Trial to Evaluate Safety, Tolerance and Pharmacokinetics of Recombinant Anti-EGFR Human Mouse Chimeric Monoclonal Antibody Injection (CDP1) in Patients With Advanced Solid Tumors
Brief Title: Phase I Clinical Trial of CDP1 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dragonboat Biopharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDP100003
Record Dates: First submitted 2019-10-29; First posted 2019-11-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Advanced Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-EGFR monoclonal antibody (Experimental): This is a dose-escalation phase, all participants will receive treatment with CDP1. Participants enrolled in this trial may receive one of the following doses dependent upon time of enrolment into the study.
  Interventions: Drug: CDP1
- anti-EGFR monoclonal antibody + chemotherapy (Experimental): This is a dose-expansion phase, participants with penile squamous cell carcinoma will receive CDP1 in combination with TIP chemotherapy.
  Interventions: Drug: CDP1; Drug: TIP chemotherapy

INTERVENTIONS:
Drug: CDP1 — Single dose part:
  Cohort 1:400 mg/m2; Cohort 2: 500 mg/m2; Cohort 3: 750 mg/m2;
  Multi-dose Part:
  Starting dose: Cohort 1:400 mg/m2; Cohort 2/3: 500 mg/m2; Maintenance dose: Cohort 1:250 mg/m2, QW; Cohort 2/3: 500 mg/m2, Q2W;
  Other Names: Recombinant anti-EGFR human mouse chimeric monoclonal antibody
  Arms: anti-EGFR monoclonal antibody
Drug: CDP1 — Starting dose: 400 mg/m2; Maintenance dose: 250 mg/m2,QW;
  Other Names: Recombinant anti-EGFR human mouse chimeric monoclonal antibody
  Arms: anti-EGFR monoclonal antibody + chemotherapy
Drug: TIP chemotherapy — Paclitaxel: 175 mg/m2 in day 1, Q3W; Ifosfamide: 1200 mg/m2 in day 1, day 2 and day 3, Q3W; Cisplatin: 25 mg/m2 in day 1, day 2 and day 3, Q3W; Participants received TIP chemotherapy up to 6 cycles (21 days per cycle).
  Arms: anti-EGFR monoclonal antibody + chemotherapy

SUMMARY:
The main purpose of this study was to evaluate the safety and tolerability of CDP1 in patients with advanced solid tumor, to explore dose limited toxicity (DLT), and to determine the recommended dose (RP2D) for phase II clinical trials.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

To evaluate the safety and tolerability of CDP1 in patients with advanced solid tumor, to explore the dose limited toxicity (DLT), and to determine the recommended dose (RP2D) for phase II clinical trial.

Secondary:

To evaluate the pharmacokinetics of CDP1 in patients with advanced solid tumor.

To evaluate the immunogenicity of CDP1 in patients with advanced solid tumor.

To evaluate the initial efficacy of CDP1 in patients with advanced solid tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 (inclusive), gender unlimited;
2. Dose-escalation phase: Patients with advanced solid tumors confirmed by histology or cytology who have failed to receive the existing standard treatment or are unable to tolerate or unwilling to accept the standard treatment (tumor types benefiting from anti EGFR treatment, including but not limited to colorectal cancer, head and neck squamous cell carcinoma, esophageal squamous cell carcinoma, penile squamous cell carcinoma, etc.); Dose-expansion phase: Patients with recurrent or metastatic advanced penile squamous cell carcinoma confirmed by histology or cytology who are not suitable for radical resection;
3. For colorectal cancer patients, RAS / BRAF was detected as wild-type.
4. ECOG physical strength score: 0-1;
5. Expected survival time over 3 months;
6. According to RECIST1.1, there is at least one tumor lesion that can be assessed;
7. No serious abnormalities of blood system, liver function, renal function and coagulation function: Neutrophils ≥1.5×10 9 /L, platelets ≥ 75 × 10 g/L, hemoglobin ≥ 90g/L;Total bilirubin ≤ 1.5ULN, ALT ≤ 2.5ULN, AST ≤ 2.5ULN (ALT ≤ 5ULN, AST ≤ 5ULN in patients with liver metastasis); Blood creatinine ≤ 1.5ULN; APTT ≤ 1.5ULN, Pt ≤ 1.5ULN, INR ≤ 1.5ULN;
8. Eligible fertile patients (male and female) must agree to use a reliable method of contraception (hormonal or barrier or abstinence) during the trial and for at least 12 weeks after the last dose; Women of childbearing age must have a negative blood or urine pregnancy test within 7 days of enrollment;
9. Subjects shall give informed consent to the study before the trial and sign written informed consent voluntarily;

Exclusion Criteria:

1. Received chemotherapy, biotherapy, radiotherapy, endocrinotherapy, small molecule targeted therapy and other anti-tumor treatment (except for nitrosourea, mitomycin C and fluorouracil oral drugs) within 4 weeks before starting to use the study drug: 6 weeks for nitrosourea or mitomycin C; The interval between the last oral administration of fluorouracil, such as tegio and capecitabine, and the use of the study drug is at least 2 weeks; Received big molecule anti-tumor drugs which had long half-lives (such as anti PD-1 or PD-L1 drugs) within 8 weeks before enrollment;
2. Received other investigational products within 4 weeks before enrollment;
3. Have received EGFR inhibitor treatment before and failed treatment;
4. Patients who have failed previous platinum therapy (Recurrent within 6 months after completion of platinum neoadjuvant/adjuvant therapy defined as treatment failure, cannot be included in this study; If the recurrence occurs after more than 6 months, the patient can be included);
5. Patients who had undergone major organ surgery (excluding puncture biopsy) or had significant trauma but not recovered within 4 weeks before admission;
6. The adverse reactions of the previous anti-tumor treatment have not been restored to CTCAE 5.0 grade evaluation ≤ 1 (except for hair loss); the radiotoxicity has not been restored to CTCAE 5.0 grade evaluation grade 1 and below (except for no effect).
7. The central nervous system metastasis without treatment or with clinical symptoms is not suitable for the group according to the judgment of the researcher; the patients suspected of brain or pia mater diseases with clinical symptoms need to be excluded by CT / MRI (flow chart notes);
8. Uncontrolled systemic infection;
9. Have a history of immunodeficiency, including HIV antibody test;
10. Treponema pallidum antibody positive;
11. Patients with chronic hepatitis B virus (HBV) infection, and the number of copies of HBV is more than 1000 IU / ml; patients with active hepatitis C virus (HCV) infection (note of index flow chart);
12. Serious cardiovascular disease history: including ventricular arrhythmia requiring clinical intervention; acute coronary syndrome, congestive heart failure, stroke or other cardiovascular events of level III and above within 6 months; NYHA heart function grade ≥ level II or left ventricular ejection fraction (LVEF) < 50%; poor control of hypertension, which is judged to be uncomfortable by researchers Join group;
13. Patients with other serious systemic diseases (including respiratory system, endocrine system, etc.) who are not suitable for clinical trials according to the judgment of researchers;
14. Known dependence on alcohol or drugs;
15. People with mental disorder or poor compliance;
16. Pregnant or lactating women;
17. In the past, when using biological products drugs, severe transfusion reaction occurred;
18. The investigator believes that the subject is not suitable for this clinical study due to any clinical or laboratory examination abnormality or other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | At the end of Cycle 1 (28 days).
  Number of participants with dose limiting toxicity (DLT)
Recommended phase II dose (RP2D) | At least one cycle of treatment(6 months).
  Recommended phase II dose (RP2D) evaluated on the first cycle.

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Observed Maximum Serum Concentration (Cmax) of CDP1 After Infusion | Up to 28 Days
  Pharmacokinetic parameters Cmax for CDP1
Pharmacokinetic Parameters: Area Under the Serum Concentration-time Curve From Time Zero to the Last Sampling Time (AUC0-t) After Infusion AUC(0-t) for CDP1 | Up to 28 Days
  AUC(0-t) for CDP1
Pharmacokinetic parameters: Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUC0-00) After Infusion Pharmacokinetic parameters: AUC(0-00) for CDP1 | Up to 28 Days
  Pharmacokinetic parameters: AUC(0-00) for CDP1
Pharmacokinetic parameters: Apparent Terminal Half-life (t1/2) of CDP1 After Infusion | Up to 28 Days
  Pharmacokinetic parameters T1/2 for CDP1
Immunogenicity indicators: Number of participants with positive anti-drug antibodies (ADA) | an average of 6 months
  Immunogenicity indicators: Number of participants with positive anti-drug
Immunogenicity indicators: Number of participants with positive neutralizing antibodies | an average of 6 months
  Immunogenicity indicators: Number of participants with positive neutralizing antibodies
Objective response rate (ORR) | an average of 6 months
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Progression-free survival (PFS) | an average of 6 months
  Progression-free survival is defined as the time from the start of treatment with CDP1 until the first documentation of disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zheng, doctor, Principal Investigator — West China Hospital
Locations (1):
- Dragonboat Biopharmaceutical,Co.,Ltd, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No